CLINICAL TRIAL: NCT05920434
Title: Gaziantep University's Clinical Research Ethics Committee
Brief Title: The Effect of Foot Reflexology and Foot Bath on Paın And Qualıty of Lıfe Applıed to Dıabetıc Neuropathıc Paın
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman Provincial Health Directorate (Other)
Responsible Party: Principal Investigator, Reva Gündoğan, Expert Nurse, Adiyaman Provincial Health Directorate
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Manuscript: NS-D-22-012
Record Dates: First submitted 2023-02-01; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Diabetic Neuropathy, Painful
Keywords: Diabetes; Neuropathic Pain; Foot Reflexology; Foot Bath
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foot reflexology group (Experimental): Individuals in the foot reflexology group were treated by the researcher once a week for a total of 60 minutes, 30 minutes on each foot, for 6 weeks (28,29) (Figure 2C).
  Interventions: Other: randomized controlled study
- Foot bath group (Experimental): In the first meeting, each participant in the foot bath group was informed about the way of doing a footbath in practice. Each participant in the foot bath group was asked to apply a foot bath for 10 minutes, 3 times a week, and twice a day for 6 weeks. A plastic foot bath tub (42 x 37 x 12 cm) without a massage function is provided for each of the participant s (Figure 2D). In order not to miss the applications, the participant was followed up by phone on the specified days (3 times a week, Monday-Wednesday-Friday). Th participant was told that the foot bath water should be at 40 degrees celsius and that his feet should be kept in water for 10 minutes, approximately 10 cm above the ankle (24). The participant came to the clinic for the forms and protective sensory examination in the 2nd, 4th, and last week.
  Interventions: Other: randomized controlled study
- Control group (No Intervention): Forms and protective sensory examination tests were applied to the participant s in the control group, as in the intervention groups, and no application was made other than standard nursing care.

INTERVENTIONS:
Other: randomized controlled study — randomized controlled study,no drugs or devices were administered to the participants.
  Arms: Foot bath group; Foot reflexology group

SUMMARY:
Introduction: Pain relief in diabetic neuropathy is one of the main goals of treatment. Foot reflexology and foot bath, which are two of the important applications of holistic approaches, reduce pain and can significantly increase the quality of life.

Objective: In the current study, it was aimed to examine the effects of foot reflexology and foot bath applied to diabetic individuals with neuropathic pain on pain and quality of life.

Method: In this randomized controlled study, the sample was randomized into three groups: (I) Foot reflexology (n: 30), (II) Foot bath (n: 30), and (III) Control (n: 30). The "Patient Information Form", "DN4 Pain Questionnaire", "Neuropathic Pain Impact on Quality-of-Life questionnaire (NePIQoL)", and "Visual Analog Scale (VAS)" were used to collect research data. In the study, a protective sensory examination was also performed with the Semmes-Weinstein Monofilament (SWM) Test and the Vibration Test (128 Hz diapason). Apart from these, foot care training was given to all patients included in the practice groups as the role of the diabetes nurse, based on the diabetic foot care training prepared by the Turkish Diabetes Association.

DETAILED DESCRIPTION:
(I) Foot reflexology group Individuals in the foot reflexology group were treated by the researcher once a week for a total of 60 minutes, 30 minutes on each foot, for 6 weeks.

(II) Foot bath group In the first meeting, each patient in the foot bath group was informed about the way of doing a footbath in practice. Each patient in the foot bath group was asked to apply a foot bath for 10 minutes, 3 times a week, and twice a day for 6 weeks. A plastic foot bath tub (42 x 37 x 12 cm) without a massage function is provided for each of the patients (Figure 2D). In order not to miss the applications, the patient was followed up by phone on the specified days (3 times a week, Monday-Wednesday-Friday). The patient was told that the foot bath water should be at 40 degrees celsius and that his feet should be kept in water for 10 minutes, approximately 10 cm above the ankle 25. The patient came to the clinic for the forms and protective sensory examination in the 2nd, 4th, and last week.

Control group Forms and protective sensory examination tests were applied to the patients in the control group, as in the intervention groups, and no application was made other than standard nursing care.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with diabetes and the value of HgbA1c ≥ 6.5,
* Participants with the DN4 ≥ 4,
* Participants with the VAS ≥ 4.

Exclusion Criteria:

* Participants who were pregnant
* Participants who received any other complementary therapy during the period of the study,
* Participants who had history of systolic blood pressure lower than 100 mmHg in the past,
* Participants who were taking systemic corticosteroids in the previous month,
* Participants who with peripheral artery disease, gonarthrosis, spinal disc herniation, ankle tendonitis, active foot ulcer, and infection
* Participants who had histories of Kidney, heart and brain diseases, rheumatic diseases, thyroid diseases, other hormonal disorders, and malignancy,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-07-19 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Pain scores | 6 weeks
  Douleur Neuropathique 4 Questions -It consists of 10 questions in total. The total scale score is calculated by giving 1 point for the yes answer given by the patient to each of the questions and examination findings, and 0 points for the no answer. The lowest score is 0, the highest 10 points can be obtained. is evaluated.
Pain severity | 6 weeks
  Visual Analog Scale (VAS)-It is an equidistant scale on a 10 cm horizontal plane, on one side of which there is no pain and on the other side the pain is "unbearable". The patient is asked to mark the point on this line that best expresses the severity of his or her pain. This distance, measured in millimeters, is interpreted as a "score" .For pain severity, 0 points are "no pain" and 10 points are "worst unbearable pain". evaluated as.

SECONDARY OUTCOMES:
Sensory level | 6 weeks
  Semmes-Weinstein Monofilament (SWM) Test-During the test, the monofilament designed to apply 10 grams of pressure to the patients is touched to the designated areas of the foot until it forms the letter C. Pressure is applied to three different areas (1st metatarsal head, plantar surface of distal hallux, 5th metatarsal plantar surface) on both feet for one second, sufficient to bend the monofilament, and patients are asked whether they feel this pressure. Expression of pressure by the patient in at least two of the three areas on the plantar surface of the foot indicates sensory loss.
Vibration sense | 6 weeks
  Vibration Test (128 Hz) diapason-It is applied to the patients in the supine position with 128 Hz Diaposan.The tuning fork is placed perpendicularly and steadily on the dorsal surface of the distal phalanx of the first toe of the foot .The felt vibration time is recorded and if the patient feels the tuning fork vibration after 10 seconds, it is considered as no vibration sense.

OTHER OUTCOMES:
The quality of life | 6 weeks
  Neuropathic Pain Impact on Quality-of-Life Questionnaire (NePIQoL)-The scale consists of 42 items in total and the item answer options are in the form of a 5-point Likert scale.Except for items 12, 15, 33, 34, which are reverse scored, all items are scored from 5-1; 5 is 'strongly agree' or 'always' and 1 is 'strongly disagree' or 'no, never'. The total score range varies between 42 and 210 .A high score on the scale indicates a low quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Reva Gundogan, Expert Nurse, Study Chair — Adıyaman Provincial Health Directorate, Adıyaman Provincial Ambulance Chief Physician
Locations (1):
- Reva Gundogan, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will be stored by researchers.

REFERENCES:
- [Background] Zakin E, Abrams R, Simpson DM. Diabetic Neuropathy. Semin Neurol. 2019 Oct;39(5):560-569. doi: 10.1055/s-0039-1688978. Epub 2019 Oct 22. PMID 31639839
- See also: Google internet link — https://pubmed.ncbi.nlm.nih.gov/31639839/